CLINICAL TRIAL: NCT07285434
Title: Clinical Study of the Therapeutic Effectiveness of In-silico-Designed, Machine Learning Inspired, and Quantum-molecularly Coupled Personalized Neoantigenic Vaccines Microlyvaq™ in Patients With Advanced Non-small Cell Lung Cancer
Acronym: Microlyvaq™
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: Biogenea Pharmaceuticals Ltd. (Industry)
Collaborators: https://interonco.gr/en/ (Unknown)
Responsible Party: Principal Investigator, John Grigoriadis PharmDrs, John Grigoriadis, PharmDr (JGrigoriadis), Principal Investigator and Chief Scientific Officer, Biogenea Pharmaceuticals Ltd.
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Biogenea2
Record Dates: First submitted 2025-11-14; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: NSCLC (Non-small Cell Lung Cancer); Squamous Lung Cancer With FGFR1 Amplification; Non-Squamous Non Small Cell Lung Cancer
Keywords: Microlyvaq™; Neoantigen vaccine; Quantum molecular coupling; AI/ML-driven personalization; Th1 polyfunctional T-cell response; Pembrolizumab combination; Circulating tumor DNA (ctDNA) monitoring
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: The Microlyvaq™ interventional study model is a non-randomized, seamless adaptive Phase II/III, histology-stratified trial in first-line advanced NSCLC. Patients are not randomized between regimens; instead, they are assigned to one of two predefined treatment arms solely on the basis of tumor histology:
  Arm 1 - Squamous NSCLC: Microlyvaq™ personalized multi-epitope vaccine administered in combination with carboplatin AUC 5, paclitaxel 175 mg/m², and pembrolizumab.
  Arm 2 - Non-squamous NSCLC: Microlyvaq™ personalized multi-epitope vaccine administered in combination with carboplatin AUC 5, pemetrexed 500 mg/m², and pembrolizumab.
  The intervention is not one-size-fits-all: within each non-randomized arm, each patient's Microlyvaq™ lot is uniquely generated using AI/ML-guided selection of neoantigens, followed by quantum molecular stability ("quantum immunogenetics") to prioritize epitopes predicted to be stably presented and highly immunogenic.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microlyvaq™ + carboplatin AUC 5, pemetrexed 500 mg/m2, pembrolizumab (Non-Squamous Backbone) (Active Comparator): Arm A: Microlyvaq™ + Carboplatin + Pemetrexed + Pembrolizumab (Non-Squamous NSCLC) Target population: Adults with advanced/metastatic non-squamous NSCLC (adenocarcinoma, large-cell, or NSCLC-NOS adjudicated non-squamous) in the first-line systemic setting, with no prior systemic therapy for metastatic disease.
  Regimen: Patients receive a personalized Microlyvaq™ multi-epitope vaccine (AI/ML- and quantum-refined, derived from tumor WES/RNA-seq and high-resolution HLA typing) administered intradermally or subcutaneously (per pharmacy manual), together with carboplatin AUC 5, pemetrexed 500 mg/m², and pembrolizumab at protocol-specified doses and schedule. Microlyvaq™ is given as a prime on Cycle 1 Day 1 (±window), with boosts around Cycle 2 (~Week 3) and Cycle 3 (~Week 6), and optional maintenance/booster doses aligned with pembrolizumab (±pemetrexed) maintenance.
  Interventions: Biological: Microlyvaq™ (Personalized Multi-Epitope Immunotherapeutic)
- Microlyvaq™ + carboplatin AUC5, paclitaxel 175 mg/m2, pembrolizumab (Squamous-Adapted Backbone) (Active Comparator): Arm A: Microlyvaq™ + carboplatin AUC5, paclitaxel 175 mg/m2, pembrolizumab (Squamous NSCLC) Target population / stratum: Adults with advanced/metastatic squamous NSCLC in the first-line systemic setting, with no prior systemic therapy for metastatic disease in this line.
  Regimen: Patients receive personalized Microlyvaq™ (AI/ML-driven epitope discovery, quantum molecular stability screening, Th1-skewed design) plus carboplatin AUC 5, paclitaxel 175 mg/m², and pembrolizumab at protocol-specified doses and schedule.
  Microlyvaq™ dosing follows the same core prime/boost structure as the non-squamous arm:
  Prime: Cycle 1 (Day 1 ± window) Boost 1: ~Week 3 (Cycle 2) Boost 2: ~Week 6 (Cycle 3) Optional continued boosters aligned with pembrolizumab maintenance. The same observation, safety, and reactogenicity monitoring rules apply as in the non-squamous arm.
  Interventions: Biological: Microlyvaq™ (Personalized Multi-Epitope Immunotherapeutic)

INTERVENTIONS:
Biological: Microlyvaq™ (Personalized Multi-Epitope Immunotherapeutic) — 1. Investigational Intervention 1.1 Microlyvaq™ (Personalized Multi-Epitope Immunotherapeutic) A patient-specific, algorithmically composed, GMP-manufactured multi-epitope immunotherapy.
  Each subject's Microlyvaq™ lot is built using:
  Whole exome sequencing (WES), RNA-seq of that subject's tumor, Matched normal DNA (when available), High-resolution HLA typing, AI/ML epitope immunogenicity ranking (tumor specificity, clonality, escape risk, Th1 bias), Quantum molecular coupling / stability modeling of peptide-HLA-TCR energetics.
  The final product intentionally contains:
  Class I-restricted epitopes (for CD8⁺ cytotoxic T cells), Class II-restricted epitopes (for CD4⁺ Th1 helper support and durability), All screened for manufacturability, sterility, and safety (GMP, QP release). Formulation / administration Multi-peptide (or peptide-adjuvant co-formulation) given intradermally/subcutaneously (route finalized in pharmacy manual).
  Co-administered with a Th1-skewing immunostimulator

SUMMARY:
Microlyvaq™ is a first-line, non-randomized, two-arm clinical trial in advanced non-small cell lung cancer (NSCLC). In both arms, patients receive a personalized multi-epitope vaccine (Microlyvaq™) on top of standard-of-care chemo-immunotherapy, with treatment tailored by histology:

Arm 1 - Squamous NSCLC: Microlyvaq™ + carboplatin AUC 5 + paclitaxel 175 mg/m² + pembrolizumab Arm 2 - Non-squamous NSCLC: Microlyvaq™ + carboplatin AUC 5 + pemetrexed 500 mg/m² + pembrolizumab Because this is a non-randomized study, patients are assigned to arms based on tumor histology (squamous vs non-squamous), not by random allocation.

The core problem it addresses is that even with pembrolizumab plus histology-appropriate chemotherapy, many patients either never respond or respond briefly and then progress. Tumors evade by exhausting T cells, excluding them from the tumor bed, evolving antigen loss, and maintaining suppressive myeloid and stromal niches. Microlyvaq™ is designed to overcome these resistance modes by actively installing new, durable, polyfunctional anti-tumor immunity rather than relying only on pre-existing T cells.

Here's how it works. Each patient's tumor is sequenced (whole exome and RNA-seq) to identify both well-known lung cancer-associated antigens (e.g. NY-ESO-1, SOX2, p53, MAGE-A4, BRAF, BMI1, FXR1, HuD, HuC, CAGE) and private neoantigens created by that tumor's specific mutations, fusions, and splice variants. From this large antigen pool, machine learning models score each candidate epitope for that specific patient. The models consider predicted HLA class I and II presentation, how efficiently the antigen will actually be processed and displayed, whether it's expressed in tumor but not healthy tissue, how essential it is to most malignant cells (to avoid easy escape), and whether it is likely to drive functional, non-exhausted T-cell responses. This is not a generic ranking; it is individualized per patient.

The most promising epitopes then undergo a quantum molecular coupling evaluation. Instead of simply asking whether a peptide binds a given HLA, Microlyvaq™ modeling simulates the peptide-MHC complex as a physical system and approximates solutions to Ĥψ = Eψ to estimate whether the peptide will form a stable, low-energy, presentation-competent conformation that a realistic T-cell receptor can dock to without high energetic penalty. Epitopes that look good in simple binding screens but are predicted to be unstable, transient, or geometrically inaccessible to TCRs are excluded. The remaining epitope set is engineered to: (1) recruit potent CD8⁺ cytotoxic T cells that can kill tumor cells, and (2) recruit CD4⁺ Th1 helper T cells that produce IFN-γ, TNF-α, and IL-2 to sustain and support those killers. The vaccine is therefore intentionally multi-epitope, Th1-biased, and patient-specific.

Each personalized Microlyvaq™ lot is manufactured under GMP and given as a prime-boost series in sync with pembrolizumab and the appropriate chemotherapy backbone for the patient's histologic arm (carboplatin/paclitaxel for squamous; carboplatin/pemetrexed for non-squamous). Timing is deliberate: chemotherapy induces immunogenic tumor cell death and antigen release and transiently "opens up" the tumor microenvironment, while pembrolizumab lifts PD-1-mediated brakes on emerging T cells. Microlyvaq™ is dosed into that vulnerable window to expand vaccine-encoded clones just as new antigen is exposed and suppression is partially relieved. The goal is to generate rapid tumor shrinkage, then sustained immune pressure on residual disease, plus epitope spreading - where the immune system begins to recognize additional tumor targets beyond those in the vaccine, making escape more difficult.

The trial itself is structured as a seamless, adaptive, non-randomized Phase I/IIa study, with two predefined histology-based arms (squamous vs non-squamous) rather than randomized treatment allocations. The primary early endpoint is objective response rate (RECIST v1.1). Key secondary endpoints include progression-free survival, duration of response, and overall survival. In addition, the study incorporates real-time translational signals as decision points, including:

1. polyfunctional Th1 and CD8⁺ responses to vaccine epitopes by ELISpot/ICS,
2. durable expansion and persistence of vaccine-linked TCR clonotypes in blood and, when feasible, in tumor,
3. rapid decline in circulating tumor DNA as an early molecular marker of tumor clearance,
4. improved tumor infiltration by CD8⁺ and Th1 cells, and
5. remodeling of the tumor microenvironment away from suppressive myeloid states. If a given histology arm shows strong clinical responses plus these immune/molecular signals, that arm can seamlessly expand into survival-powered confirmation. If it does not, predefined futility rules allow that arm to stop, all within this non-randomized, adaptive framework.

DETAILED DESCRIPTION:
This is an early Phase I, non-randomized, open-label, histology-stratified, two-arm interventional study evaluating Microlyvaq™, a personalized multi-epitope peptide vaccine, in combination with first-line pembrolizumab and platinum-based chemotherapy in adults with advanced or metastatic non-small cell lung cancer (NSCLC).

Patients are assigned to treatment arm according to tumor histology only (no randomization):

* Arm 1 (Squamous NSCLC): Microlyvaq™ + carboplatin AUC 5 + paclitaxel 175 mg/m² + pembrolizumab.
* Arm 2 (Non-squamous NSCLC): Microlyvaq™ + carboplatin AUC 5 + pemetrexed 500 mg/m² + pembrolizumab, with standard folate, vitamin B12, and corticosteroid premedication.

Rationale and Unmet Need Pembrolizumab plus platinum-based chemotherapy is a standard first-line option in metastatic NSCLC and improves survival compared with chemotherapy alone. However, many patients never respond, and responders often experience early progression. Current biomarkers (e.g., PD-L1 expression or tumor mutational burden) do not reliably predict durable benefit. Major causes of failure include incomplete or exhausted tumor-reactive T-cell repertoires, stromal and vascular barriers to T-cell infiltration, immunosuppressive myeloid and cytokine milieus, metabolic constraints in the tumor microenvironment, and antigenic escape under immune pressure. Releasing PD-1-mediated inhibition, even together with chemotherapy-induced antigen release, often does not generate a sustained, diversified, polyfunctional anti-tumor immune response.

Microlyvaq™ is designed to introduce into each patient a de novo, computationally defined set of tumor-directed T-cell specificities that are tailored to the individual tumor mutational and antigenic landscape, aligned with the patient's HLA genotype, and biased toward clonally important, difficult-to-lose lesions to reduce antigen-loss escape. The vaccine is administered in a prime-boost schedule intentionally synchronized with pembrolizumab and the histology-appropriate chemotherapy backbone.

The overarching early Phase I hypothesis is that a personalized multi-epitope vaccine can be safely integrated with standard chemo-immunotherapy, will induce measurable polyfunctional T-cell responses and favorable biomarker changes, and may provide preliminary signals of deeper and more durable clinical responses than would be expected with chemo-immunotherapy alone, thereby justifying later-phase studies.

Microlyvaq™ Platform (Tumor Profiling and Epitope Selection) For each participant, tumor material is analyzed using next-generation sequencing and HLA typing to generate a patient-specific pool of candidate antigens, including private neoantigens (from non-synonymous mutations, indels, fusions or splice variants) and selected tumor-associated antigens that are overexpressed in NSCLC. An AI/machine-learning-based immunogenetic scoring system evaluates each candidate epitope with respect to predicted HLA binding, processing and presentation, tumor specificity, clonality, and likelihood of immune escape. Quantum-inspired structural modeling is then used to further prioritize peptides predicted to form stable peptide-MHC complexes that are accessible to T-cell receptors. From this process, a finite panel of class I and class II peptides is selected to compose the personalized Microlyvaq™ lot for that patient.

The epitope selection algorithm is "context-aware" of the planned chemotherapy backbone (carboplatin/paclitaxel in Arm 1 vs carboplatin/pemetrexed in Arm 2), recognizing that these regimens differentially shape patterns of tumor cell death, vascular and stromal remodeling, and transient changes in lymphoid and myeloid compartments. Panels are therefore optimized with respect to both the patient's tumor biology and the expected treatment-induced immune milieu.

Manufacturing and Administration Microlyvaq™ is manufactured under Good Manufacturing Practice (GMP) conditions. Selected peptides are synthesized, purified, and blended into a multi-epitope peptide formulation, with standard identity, purity, sterility, and endotoxin testing and verification of chain-of-identity and chain-of-custody. Feasibility endpoints include the proportion of enrolled patients in whom a Microlyvaq™ lot can be successfully generated and released within a clinically relevant time window from biopsy to first vaccination, as well as logistical performance across manufacturing, storage, shipping, and on-site handling.

The vaccine is administered by subcutaneous or intradermal injection (final route defined in the protocol) in a prime-boost schedule coordinated with pembrolizumab and chemotherapy (e.g., a prime in Cycle 1 followed by boosts in subsequent cycles and, where appropriate, during pembrolizumab maintenance). Standard premedication and post-dose observation are used to monitor for local and systemic reactions.

Study Objectives and Assessments Because this is an early Phase I non-randomized trial, the primary focus is on safety, tolerability, and feasibility of integrating Microlyvaq™ into standard first-line regimens for squamous and non-squamous NSCLC. Treatment-emergent adverse events, serious adverse events, and immune-related adverse events will be collected and graded using standard criteria. Feasibility measures include adherence to the planned vaccination schedule and the ability to deliver individualized vaccine lots on time.

Key secondary and exploratory objectives include evaluation of vaccine-induced CD4⁺ and CD8⁺ T-cell responses against vaccine-encoded epitopes, T-cell receptor (TCR) repertoire dynamics (clonal expansion and persistence of vaccine-linked clonotypes), circulating tumor DNA (ctDNA) kinetics, and changes in the tumor microenvironment in patients who consent to on-treatment biopsies. Preliminary anti-tumor activity (e.g., overall response rate, duration of response, progression-free survival and overall survival per RECIST v1.1) will be described separately in each arm; the study is not powered for formal inter-arm comparisons.

Patient Population and Treatment Eligible patients are adults with advanced (stage IIIB/IIIC) or metastatic (stage IV) NSCLC who are candidates for first-line pembrolizumab plus platinum-based chemotherapy according to local standards, have ECOG performance status 0-1, adequate organ function, and sufficient tumor tissue for sequencing and HLA typing. Patients with squamous histology are assigned to Arm 1; those with non-squamous histology (e.g., adenocarcinoma or large-cell) are assigned to Arm 2. Key exclusions include prior PD-1/PD-L1/CTLA-4 blockade in the metastatic setting, uncontrolled CNS metastases, and clinically significant active autoimmune disease. Full eligibility criteria are specified elsewhere in the protocol.

Safety Monitoring and Oversight Patients will undergo regular clinical evaluations, laboratory testing, and radiologic assessments. Dosing of Microlyvaq™, pembrolizumab, and chemotherapy may be withheld, modified, or discontinued according to protocol-defined criteria in the event of toxicity. Immune-related toxicities will be managed in accordance with contemporary guidelines for checkpoint inhibitors, with additional guidance for suspected vaccine-related events. An independent Data Safety Monitoring Board (DSMB) will periodically review accumulating safety, feasibility, and emerging efficacy/biomarker data and may recommend modification, temporary suspension, or early termination of one or both histology-defined arms if warranted.

Sample Size and Design Summary The initial safety cohort will enroll 12 patients who will be evaluable for toxicity. If no Microlyvaq™-related adverse event of > Grade 2 is observed in more than 3 patients and no Grade 4 Microlyvaq™-related toxicity is observed in any patient, enrollment may expand to a total of 30 patients across both non-randomized arms. Data from this early Phase I study are intended to support the feasibility, safety, and biological activity of Microlyvaq™ and to guide the design of subsequent Phase Ib/II trials in squamous and non-squamous NSCLC.

ELIGIBILITY:
Inclusion Criteria:

-

Subjects are eligible if all of the following are met:

Age

≥18 years at the time of informed consent. Diagnosis / Histology

Histologically or cytologically confirmed non-small cell lung cancer (NSCLC) that is:

Non-squamous (e.g. adenocarcinoma, large-cell, NSCLC-NOS adjudicated non-squamous), or Squamous (if/when that stratum is open). Diagnosis must be locally documented and source-verifiable. Stage / Disease Status Stage IIIB / IIIC / IV or recurrent/metastatic NSCLC not amenable to curative surgery or radiotherapy, per AJCC 8th edition staging.

Disease is considered first-line metastatic/systemic setting:

No prior systemic therapy for advanced/metastatic disease in this line. Prior adjuvant/neoadjuvant therapy or consolidation chemo-RT is allowed if completed and the subject relapsed outside the protocol-defined disease-free interval (e.g. relapse ≥6-12 months after completion, per final protocol text).

Measurable Disease At least one measurable lesion per RECIST v1.1 at baseline imaging. Baseline imaging must be within 28 days prior to Day 1 (CT chest/abdomen/pelvis ± contrast, plus brain MRI if clinically indicated).

ECOG Performance Status ECOG 0 or 1 at screening. Subject must be ambulatory and clinically stable enough to receive combination therapy (pembrolizumab + chemo ± Microlyvaq™).

Adequate Organ and Marrow Function (Representative thresholds - to be finalized numerically in the protocol SOP, but typically:) Absolute neutrophil count (ANC) ≥1.5 × 10⁹/L. Platelets ≥100 × 10⁹/L. Hemoglobin ≥9.0 g/dL (transfusion allowed per institutional standard prior to enrollment).

AST and ALT ≤2.5 × upper limit of normal (ULN), or ≤5 × ULN if liver metastases are present.

Total bilirubin ≤1.5 × ULN (≤3 × ULN if known Gilbert's syndrome). Creatinine clearance / eGFR ≥45 mL/min/1.73 m² (sufficient for pemetrexed/platinum; final numeric cutoff may align to pemetrexed label).

Coagulation: INR and aPTT compatible with safe biopsy (if biopsy expected) per site policy.

Oxygenation: No resting hypoxemia prohibitive for safe treatment in investigator judgment.

Tumor Tissue Availability

Adequate tumor material must be available for:

PD-L1 assessment, DNA/RNA extraction (whole exome sequencing / RNA-seq or targeted panel sufficient for epitope discovery), High-resolution HLA typing support, Optional spatial profiling.

Acceptable sources:

Recent core needle biopsy or surgical specimen (preferred), OR Archival FFPE block or ≥15 unstained slides with documented tumor cellularity. Tumor cellularity must meet the minimum input requirement for sequencing and PD-L1 scoring (macrodissection allowed).

Biospecimen / Translational Willingness

Willing and able to provide required blood samples at protocol-defined timepoints:

PBMC (for ELISpot, ICS, TCR sequencing), Plasma/serum (for ctDNA, exosomal miRNA, cytokines), HLA typing. Willing to allow shipment of these biospecimens under chain-of-custody to central labs.

Willing to undergo optional on-treatment biopsy (e.g. around Cycle 3 / ~Week 6-9) if, in the investigator's judgment, it is clinically safe and technically feasible. If unsafe, liquid biopsy alone is acceptable.

Contraception / Reproductive Status Females of childbearing potential: negative pregnancy test at screening and prior to first dose.

Females of childbearing potential and males with partners of childbearing potential must agree to use highly effective contraception during study treatment and for the protocol-defined post-treatment window:

Typically ≥120 days after last pembrolizumab dose and ≥90 days after last Microlyvaq™ dose, whichever is longer (final timing per protocol).

No intention to conceive or donate gametes during this protection window. Informed Consent

Capable of understanding and signing informed consent(s), including:

Main study consent (chemo + pembrolizumab + Microlyvaq™), Genomic profiling / HLA typing consent, Optional on-treatment biopsy / leukapheresis consent (if applicable at site), Data/privacy language (GDPR-compliant). Willing to comply with study visits, dosing schedule, safety monitoring, PRO questionnaires (if enrolled in PRO subset), and survival follow-up.

Exclusion Criteria:

Subjects must not meet any of the following:

Prior Systemic Therapy in Metastatic Setting Any prior systemic therapy for metastatic / unresectable NSCLC in the current line.

Exception: prior adjuvant/neoadjuvant chemo, IO, or chemoradiation allowed if relapse occurred outside the protocol's defined exclusion interval (e.g. relapse ≥6-12 months after completion); exact interval to be specified.

Known Oncogene-Addicted Disease Requiring Targeted SOC Subjects whose tumors harbor actionable drivers for which an approved targeted therapy is standard first-line care (e.g. EGFR activating mutation, ALK rearrangement, ROS1 rearrangement, certain ERBB2/HER2 drivers, MET exon 14 skipping, RET fusion, NTRK fusion, KRAS G12C where local standard is targeted frontline) may be excluded or enrolled only in specific sub-cohorts if allowed by the statistical design.

Rationale: It may be unethical to withhold proven first-line targeted agents. The final protocol will define whether these genotypes are (a) excluded, (b) stratified, or (c) routed to a molecularly restricted exploratory cohort.

Uncontrolled CNS Disease Active, symptomatic brain metastases or leptomeningeal disease requiring immediate local intervention.

Allowed:

Previously treated/stable brain metastases are permitted if:

Clinically stable, Off high-dose steroids (e.g. >10 mg prednisone equivalent daily) for ≥14 days before Day 1, No new/worsening neurologic symptoms for ≥2 weeks.

Excluded:

Ongoing steroid dependency above immunosuppressive thresholds, uncontrolled seizures, mass effect with high intracranial pressure, or unstable neuro deficits judged unsafe.

Autoimmune / Immune-Mediated Conditions of Concern Active, uncontrolled autoimmune disease that has required systemic immunosuppression >10 mg/day prednisone-equivalent (or biologic immunosuppressive agent) within 14 days prior to Day 1.

History of severe (life-threatening) immune-related adverse event (irAE) to prior PD-1/PD-L1/CTLA-4 (e.g. Grade 4 pneumonitis, myocarditis, neurologic irAE that did not fully resolve), unless cleared by Medical Monitor.

Autoimmune disorders that are mild, stable, and not expected to flare under PD-1 blockade (e.g. controlled hypothyroidism on replacement; vitiligo; stable type 1 diabetes on insulin) may be allowed.

Significant Active Infection Any uncontrolled active infection requiring IV antibiotics or hospitalization at screening.

Uncontrolled HBV, HCV, or HIV viremia above protocol thresholds:

HBV: high viral load without appropriate antiviral management. HCV: untreated, high-level viremia with ongoing hepatic decompensation. HIV: uncontrolled (e.g. not on stable antiretroviral therapy, CD4 below a prespecified safe cutoff); final numeric cutoffs defined in protocol.

Active tuberculosis or other serious opportunistic infection. Clinically Significant Pulmonary Compromise Baseline pneumonitis requiring steroids. Prior ≥Grade 3 immune-mediated pneumonitis from checkpoint inhibitor therapy that did not resolve to ≤Grade 1.

Severe, uncontrolled interstitial lung disease that would make pembrolizumab plus investigational immunostimulation unsafe.

Other Serious Uncontrolled Comorbidities Uncontrolled congestive heart failure, unstable angina, recent myocardial infarction or stroke (typically <6 months).

Clinically significant uncontrolled arrhythmia. Severe uncontrolled hypertension. Any condition that, in the investigator's judgment, would make study therapy unacceptably high risk (e.g. ECOG drift, frailty, severe malnutrition).

Bleeding Risk / Biopsy Unsuitability (When Biopsy is Expected) Active, clinically significant bleeding or coagulopathy that cannot be corrected.

Platelet count or anticoagulation status that, in investigator judgment, makes mandatory biopsy unsafe.

NOTE: If a site/arm requires an on-treatment biopsy for core analysis and it is deemed unsafe, subject may still be eligible if protocol allows liquid-biopsy-only participation in that stratum. (This must be explicitly permitted to avoid excluding medically fragile patients.) Known Hypersensitivity Known severe hypersensitivity (e.g. anaphylaxis) to pembrolizumab, to the planned chemotherapy backbone (e.g. pemetrexed, carboplatin) despite standard premedication strategies, or to critical Microlyvaq™ excipients / adjuvant components.

In pemetrexed-containing regimens: inability/unwillingness to receive mandatory folate and vitamin B12 supplementation and steroid premedication.

In carboplatin regimens: uncontrolled prior carboplatin hypersensitivity not manageable by desensitization.

Pregnancy / Breastfeeding Pregnant or breastfeeding at screening. Intention to become pregnant (or impregnate a partner) during study therapy or within the required contraception window after last dose.

Concurrent Participation in Confounding Interventional Trials Enrollment in another interventional clinical study that could confound efficacy/safety readouts or interfere with immune profiling.

Exceptions:

Non-interventional / observational registries, Certain supportive care trials with Medical Monitor approval, Protocol-approved combination substudies (if integrated under the Microlyvaq™ umbrella and statistically planned).

Any Condition That Interferes With Protocol Compliance

Inability or unwillingness to comply with:

Scheduled visits, Biospecimen collections (for HLA typing, PBMC isolation, ctDNA, etc.), Imaging schedule (q6 weeks through Week 24, then q9-12 weeks), Safety follow-up and PRO questionnaires (if PRO subset), Survival follow-up calls ~q12 weeks post-treatment. Cognitive, psychiatric, or social situations that in the investigator's judgment would preclude safe, reliable participation and follow-up.

Notes / Operational Clarifiers

HLA typing and sequencing feasibility:

The subject must have enough viable tumor + PBMC DNA/RNA to allow:

WES / RNA-seq or equivalent targeted sequencing for neoantigen discovery, High-resolution HLA-A/B/C typing. If a subject cannot generate a viable personalized epitope set (e.g. insufficient material for immunogen design), that subject may be ineligible for Microlyvaq™ dosing but could be eligible for safety follow-up / SOC reference cohorts, depending on how the arm is structured.

Brain metastases:

Stable, treated, asymptomatic brain mets are allowed. This matters in first-line metastatic NSCLC, because excluding all brain mets would make the trial clinically irrelevant. The key exclusion is uncontrolled CNS disease requiring urgent steroids/radiation/surgery.

Actionable oncogene drivers:

Final protocol must say explicitly whether EGFR/ALK/ROS1/etc. are:

excluded entirely, allowed but stratified, or diverted to exploratory "post-standard-targeted-therapy" cohorts. This is both ethical and regulatory: you don't want to randomize someone away from globally recognized, mutation-directed SOC.

Autoimmune disease:

The bar is not "no autoimmune history ever." It's "no uncontrolled, high-risk autoimmune activity that would likely flare catastrophically when we give a personalized Th1-skewing vaccine + PD-1 blockade."

Contraception window:

Needs to line up with pembrolizumab label and with any reproductive toxicity data from Microlyvaq™ (e.g. ≥120 days / ≥90 days windows). Keep that harmonized across patient materials, pharmacy manual, and consent.

This criteria block is inspection-facing: it protects safety, preserves interpretability of immune endpoints, ensures we can actually manufacture/deliver a personalized Microlyvaq™ lot, and keeps the population consistent with first-line pembrolizumab+chemo standards in advanced NSCLC.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2028-02-02 (Estimated); Study Completion 2030-02-02 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS): AI epitope ranking, quantum energetics, TCR repertoire engineering, ctDNA collapse, spatial immune remodeling - is in service of extending OS safely. Subjects alive at cut-off are censored at last known alive. | Survival status assessed approximately every 12 weeks during long-term follow-up, through study completion, up to approximately 36 months.
  Overall survival is the time from first dose of study treatment to death from any cause. Survival will be summarized with Kaplan-Meier curves; between-arm comparisons will use a stratified Cox model to estimate hazard ratios (HRs) with 95% confidence intervals (CIs). If non-proportional hazards are detected, restricted mean survival time (RMST) will be used. Stratification factors may include PD-L1 proportion score (TPS), smoking status, actionable driver status (EGFR/ALK/ROS1/ERBB2/KRAS-G12C), and geographic region. Subsequent anti-cancer therapy after progression will not reset survival time (treatment-policy strategy). Patients lost to follow-up will be censored at the last date known alive. Overall survival will be evaluated in two non-randomized histology cohorts: Arm 1 (squamous NSCLC): Microlyvaq™ + carboplatin + paclitaxel + pembrolizumab; Arm 2 (non-squamous NSCLC): Microlyvaq™ + carboplatin + pemetrexed + pembrolizumab (with folate/B12 and steroid support).
Objective Response Rate (ORR; Confirmed CR+PR): The Microlyvaq™ vaccine is delivered into a "window of susceptibility": right when chemotherapy has induced immunogenic cell death and pembrolizumab has lifted PD-1 brakes on on exhausted T cells. | Confirmation window: Response must be confirmed 8 weeks after first CR/PR call, so typically ~Week 14 for first responders.Update cadence: Every imaging timepoint: 6 weeks through Week 24, then 12 weeks thereafter.
  * ORR (%) with 95% CI in the Full Analysis Set (all randomized with measurable disease at baseline).
  * Between-arm comparison via stratified CMH or logistic regression adjusting for prespecified strata.
  * Missing confirmatory scan defaults to "non-responder" in the primary analysis to avoid false inflation.
  In Microlyvaq™, ORR is not just "does tumor shrink." It's "does our AI / ML / quantum-informed control signal actually force the tumor-immune system into the kill state we predicted, on schedule."• Each Microlyvaq™ lot is not a fixed commercial SKU. It's a computationally composed payload of ~17-25 epitopes, each picked for that exact patient by AI/ML plus quantum energy modeling to maximize productive peptide-HLA display, stable TCR engagement geometry, and resistance to tumor immune escape. In Microlyvaq™, ORR is not just "does tumor shrink." It's "does our AI / ML / quantum-informed signal actually force the tumor-immune system into the kill state we predicted, on schedule"

SECONDARY OUTCOMES:
Progression-Free Survival (PFS): Time from randomization to first of either: 1. RECIST v1.1 progression (investigator), or 2. Death from any cause. Sensitivity analysis uses blinded ERC progression calls. | Time Frame: From baseline (scan within 28 days before Day 1) through study completion, with tumor assessments every 6 weeks through Week 24, then every 12 weeks thereafter (up to approximately 24 months).
  * Kaplan-Meier curves, stratified log-rank test, and stratified Cox HR with 95% CI.
  * Handling of new therapy before documented PD: in the primary analysis, switching early to another systemic therapy is treated as if progression occurred at the last adequate tumor assessment; sensitivity analysis censors at switch and relies on ERC adjudication.
  If PFS meaningfully improves and aligns with immune readouts (ctDNA suppression, sustained TCR clones, maintained intratumoral CD8⁺/Th1 infiltration), that's strong mechanistic validation. PFS measures whether the new immune repertoire we engineered (Th1-supported, polyfunctional, persistent TCR clonotypes) is actually able to hold the tumor in a suppressed state under real-world stress - metabolic starvation, stromal exclusion, myeloid suppression, spatial heterogeneity - once the initial cytotoxic wave is over.
Duration of Response (DoR) for confirmed responders (CR/PR) | From end of on-treatment follow-up, survival status assessed approximately every 12 weeks through study completion, up to approximately 36 months.
  Duration of response (DoR) is defined, for participants with confirmed complete or partial response (CR/PR), as the time from first documented response to RECIST v1.1 progression or death; participants without an event are censored at the last adequate tumor assessment. DoR will be summarized using Kaplan-Meier curves in responders, with median DoR and 95% confidence intervals, and sensitivity analyses using independent ERC review and alternative censoring at the start of new anti-cancer therapy. Exploratory analyses may overlay ctDNA kinetics during DoR to show molecular durability alongside radiologic durability, as a readout of persistence of vaccine-induced T-cell responses and the underlying epitope-selection strategy.
Disease Control Rate (DCR): CR + PR + durable stable disease (SD ≥6 weeks at the first scheduled post-baseline scan). | From the first post-baseline tumor assessment (approximately Week 6) through confirmation of disease control, with tumor assessments every 6 weeks through Week 24, then every 12 weeks thereafter through study completion (up to approximately 24
  Disease Control Rate (DCR): Proportion of patients with complete response (CR), partial response (PR), or stable disease (SD) lasting ≥ 6 weeks at or beyond the first scheduled post-baseline tumor assessment, per RECIST v1.1. In metastatic NSCLC, DCR captures not only overt tumor shrinkage but also durable "immune-mediated stalemate," where Microlyvaq™ may convert immune-cold, myeloid-rich lesions into inflamed, T-cell-infiltrated tumors that stop progressing but do not fully regress.
  Analysis: Proportion (with 95% confidence interval) in the full analysis set with measurable disease; between-arm comparisons using logistic regression and/or Cochran-Mantel-Haenszel (CMH) methods stratified by prespecified factors.
Time to Response (TTR):Among responders, time from randomization to first confirmed CR/PR. | First evaluable: First scan with CR/PR (~Week 6).Confirmation anchor: Responses are only counted once confirmed 4-8 weeks later (so confirmed TTR for early responders ~Week 10-14).
  The Microlyvaq™ prime/boost schedule is phase-matched to chemo/pembro timing windows when antigen release, checkpoint relief, and vascular access are maximized. If we got the timing right, responses shouldn't be mysteriously delayed; they should start to appear in those synchronized windows. A long lag with late "catch-up" responses might signal mis-phasing of u(t).
  * Median TTR and distribution descriptions across arms.
  * Non-parametric comparisons with caveats about responder-only bias.
Incidence of Treatment-Emergent Adverse Events (TEAEs) | From first dose of any study drug through 30 days after the last dose of any study drug (up to approximately 12 months, depending on treatment duration).
  Incidence, severity, and relationship to study treatment will be summarized by arm for all treatment-emergent adverse events (TEAEs), including Grade ≥3 TEAEs and TEAEs leading to treatment discontinuation. By-arm incidence tables and exposure-adjusted incidence rates will be presented. A narrative review will be provided for any severe systemic inflammatory TEAEs temporally associated with Microlyvaq™.
Time to Sustained Deterioration in LC13 Lung Symptoms (Dyspnea, Cough, Chest Pain) | From baseline (Day 1) until the first sustained deterioration in LC13 score or death, whichever occurs first, assessed up to approximately 24 months.
  Time from baseline to the first ≥10-point worsening from baseline in prespecified EORTC QLQ-LC13 lung symptom items (dyspnea, cough, chest pain) that is confirmed (i.e., persists) at the next scheduled assessment; death before the next assessment is counted as deterioration in the primary analysis. This endpoint evaluates whether treatment delays clinically meaningful worsening of lung symptoms (patients breathing better, coughing less, and having less chest pain). Time to deterioration will be analyzed using Kaplan-Meier methods with stratified Cox hazard ratios and 95% confidence intervals; mixed models for repeated measures (MMRM) will be used to describe mean symptom changes over time as supportive analyses.

OTHER OUTCOMES:
Incidence of Procedure-Related Serious Adverse Events (SAEs) | From baseline (Day 1) through study completion, up to approximately 36 months.
  Percentage of participants with ≥1 serious adverse event judged related to protocol-mandated procedures (e.g., tumor biopsies, leukapheresis), such as bleeding, pneumothorax, sepsis, or hemodynamic instability. Events will be coded using MedDRA and summarized descriptively, with the primary reported value being the proportion of participants experiencing at least one procedure-related SAE.
Change From Baseline in EORTC QLQ-C30 Global Health Status/Quality of Life (QoL) Score | From baseline (Day 1) through end of study or up to approximately 36 months, with EORTC QLQ-C30 assessments collected at scheduled study visits (approximately every 3 weeks through Week 24, then every 9-12 weeks thereafter).
  Change from baseline in the EORTC QLQ-C30 global health status/QoL score will be assessed over time; mean change from baseline and the proportion of participants with a clinically meaningful change (≥10-point improvement or worsening) will be reported. Analysis will use a mixed model for repeated measures (MMRM) with fixed effects for treatment, time, treatment-by-time interaction, and baseline score.
Proportion of Patients Achieving ctDNA Major Molecular Response (MMR) | From baseline (pre-treatment sample) to the first on-treatment ctDNA assessment at approximately Week 6 (with an assessment window extending up to Week 9).
  ctDNA MMR is defined as a predefined large reduction (e.g., ≥80-90%) from baseline in circulating tumor DNA variant allele fraction for patient-specific driver or truncal variants at the first on-treatment landmark. The primary reported value is the proportion of patients with ctDNA MMR; exploratory analyses will assess associations between ctDNA MMR and objective response rate (ORR), progression-free survival (PFS), and overall survival (OS).
Vaccine-Linked TCR Clonotype Expansion and Persistence | From baseline (pre-vaccination) through post-vaccination landmark assessments at approximately Week 6, Week 13, Week 25, and up to 90 days after the last immune-active dose.
  Change from baseline in the frequency of T-cell receptor (TCR) clonotypes specific for Microlyvaq™-selected epitopes will be quantified in peripheral blood (and, where available, tumor tissue). The reported value will be the fold-change from baseline in vaccine-linked clonotype abundance at predefined post-vaccination landmark time points.
Change From Baseline in Polyfunctional Th1/Cytotoxic T-Cell Responses (ELISpot/ICS) | Baseline (Day 1, pre-vaccination) and approximately Week 13 after start of treatment.
  Change from baseline in the frequency (percentage) of antigen-specific T cells producing multiple Th1/cytotoxic cytokines (e.g., IFN-γ, TNF-α, IL-2, with or without granzyme/perforin) upon ex vivo restimulation with Microlyvaq™-selected epitopes, as measured by ELISpot and/or intracellular cytokine staining (ICS). The reported value will be the mean (and/or median) change from baseline in polyfunctional T-cell frequency, reflecting vaccine-induced Th1/cytotoxic immune activation.
Change From Baseline in Intratumoral CD8⁺ T-Cell Density | Baseline (pre-treatment, Day 1) and on-treatment biopsy at approximately Week 13 after start of study therapy.
  Change from baseline in intratumoral CD8⁺ T-cell density (within tumor nests) between baseline and on-treatment biopsies. The reported value will be the mean (and/or median) change from baseline in CD8⁺ T-cell density, reflecting increased intratumoral T-cell infiltration.

CONTACTS AND LOCATIONS:
Locations (1):
- Biogenea Pharmaceuticals Ltd, Thessaloniki, Macedonia, Greece

IPD SHARING:
Plan to Share IPD: Yes
The following de-identified, participant-level data will be included:
  Core clinical efficacy data Demographics and baseline disease characteristics (e.g. age, sex, ECOG performance status, histology, PD-L1 tumor proportion score strata, presence/absence of actionable oncogenic drivers).
  Treatment assignment (study arm) and treatment exposure (dates and number of cycles of Microlyvaq™, pembrolizumab, platinum/taxane or pemetrexed-based chemotherapy).
  Tumor response assessments per RECIST v1.1 (target lesion measurements, best overall response, confirmation status).
  Time-to-event endpoints: progression-free survival (PFS), duration of response (DoR), overall survival (OS), and censoring information (dates and reasons).
  Disease control status at protocol-defined timepoints. Concomitant anti-cancer therapies received after on-study treatment discontinuation.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The IPD package described above will be prepared after:
  Database lock for the primary clinical analysis of the relevant cohort/arm, Resolution of all serious safety queries for that analysis set, Acceptance or public presentation/publication of primary efficacy and key safety results.
  A structured dictionary / codebook (variable definitions, derivations, censoring rules) will accompany the shared IPD so that outside investigators can interpret the fields without needing access to internal SOPs.
Access Criteria: We will share de-identified, subject-level clinical efficacy, safety, imaging-derived response calls, ctDNA kinetics summaries, T-cell pharmacodynamic summaries (polyfunctionality and clonal expansion/persistence scores), and predefined tumor microenvironment scores. We will not broadly release raw genomic sequences, raw TCR sequences, full unmasked pathology images, or any directly identifying information. Access to more granular molecular data can be requested, but will require enhanced review, additional agreements, and documented safeguards.
URL: https://myoncotherapy.com